CLINICAL TRIAL: NCT03664661
Title: a Single-center, One Arm, Open Clinical Study of BCMA Nanobody CAR-T Cell in Refractory/Relapsed Myeloma
Brief Title: BCMA-CAR-T in Relapsed/Refractory Multiple Myeloma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: The Pregene (ShenZhen) Biotechnology Company, Ltd. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HenanCH CAR 2-2
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Relapsed/Refractory Myeloma
MeSH Terms: conditions — Neoplasms, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): BCMA nanobody CAR-T cells
  Interventions: Drug: BCMA nanobody CAR-T cells

INTERVENTIONS:
Drug: BCMA nanobody CAR-T cells — step 1: Collect 50-100ml of peripheral blood for culture of BCMA nanobody CAR- T cells. step 2. After 72 hours, pretreated with FC regimen, details as follow Cyclophosphamide 600-800mg/m2 for 2 days Fludarabine 25-30mg/m2 for 3 days. step 3: After another 48 hours transfusion the cells back to the patients the numbers of infused CAR T cells are 5x106 /kg for the first 3 patients, 1.5x107 /kg for the second 3 patients and 4.5x107 /kg for the third 3 patients.
  After finishing this, another 6 patients will be enrolled for observation of efficacy.

SUMMARY:
Evaluation of the safety and efficacy of BCMA nanobody CAR-T cells in relapsed/refractory myeloma

DETAILED DESCRIPTION:
There are no effective regimens for relapsed/refractory myeloma. BCMA express extensively in mature B cells and plasma cells. Myeloma cells express BCMA universally. BCMA signal pathway can induce plasma cell proliferation and survival, down-regulation of BCMA could control the progression of myeloma. The BCMA CAR used in this study consists of BCMA nanobody, CD8 hinge, transmembrane region and 4-1bb co-stimulation domain.

ELIGIBILITY:
Inclusion Criteria:

* 18 and ≤70 years old and the expected lifetime >3 months

  * Active myeloma according to IMWG criteria, and BCMA positive by immunohistochemistry or flow cytometry
  * No effective treatment option available
  * ECOG score 0-2
  * Sufficient heart, liver, kidney function (heart: no heart disease or coronary heart disease, patient heart function NYHA grade 1-2; liver: TBIL ≤ 3ULN, AST ≤ 2.5ULN, ALT ≤ 2.5ULN; kidney: Cr≤ 1.25ULN);
  * smoothly peripheral superficial veins
  * No other serious diseases that conflict with this protocol (eg, autoimmune diseases, immunodeficiency, organ transplantation)
  * No history of other malignancies
  * Women of childbearing age must be negative for blood pregnancy test within 7 days and must take appropriated contraceptive measures during and 3 months after the study
  * The patient himself agrees to participate in this clinical study and signed the "informed consent"

Exclusion Criteria:

* Severe infectious 4 weeks before enrollment
* Active hepatitis B or C viral hepatitis, HIV,
* Severe autoimmune disease or immunodeficiency disease
* Severe allergies
* Severe mental disorder
* Patients who used high-dose glucocorticoids within 1 week
* Participation in other clinical studies in the past 3 months or having been treated with other gene products

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-04-11 (Actual); Primary Completion 2019-04-10 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
occurrence of study related adverse events | 4 weeks
  safety of CAR-T cells

SECONDARY OUTCOMES:
Treatment response rate | 3 months and 6 months
  response rate according to IMWG criteria
copy number of CAR-T cells | one year
  copy number of CAR-T cells

CONTACTS AND LOCATIONS:
Overall Officials: Yongping Song, M.D, Study Chair — Henan Cancer Hospital
Locations (1):
- Cancer Hospital Affiliate to Zhengzhou University & Henan Cancer Hospital, Zhengzhou, Henan, China